CLINICAL TRIAL: NCT04785287
Title: Phase I/II Trial of Anti-CTLA4-NF mAb (BMS-986218) in Combination With Nivolumab and Hypofractionated Stereotactic Radiation Therapy in Patients With Advanced Solid Malignancies
Brief Title: Anti-CTLA4-NF mAb (BMS986218), Nivolumab, and Stereotactic Body Radiation Therapy for the Treatment of Metastatic Solid Malignancies
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2020-0479; NCI-2021-01619 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2020-0479 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2021-03-04; First posted 2021-03-05 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Advanced Lung Carcinoma; Advanced Malignant Solid Neoplasm; Malignant Adrenal Gland Neoplasm; Metastatic Liver Carcinoma; Metastatic Lung Carcinoma; Metastatic Malignant Solid Neoplasm; Stage III Liver Cancer; Stage III Lung Cancer AJCC v8; Stage IIIA Lung Cancer AJCC v8; Stage IIIB Lung Cancer AJCC v8; Stage IIIC Lung Cancer AJCC v8; Stage IV Liver Cancer; Stage IV Lung Cancer AJCC v8; Stage IVA Liver Cancer; Stage IVA Lung Cancer AJCC v8; Stage IVB Liver Cancer; Stage IVB Lung Cancer AJCC v8
MeSH Terms: conditions — Adrenal Gland Neoplasms; Carcinoma, Hepatocellular; Lung Neoplasms; Neoplasm Metastasis; Liver Neoplasms | interventions — Nivolumab; Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm I (BMS-986218, SBRT) (Experimental): Patients receive anti-CTLA4 monoclonal antibody BMS-986218 IV over 30 minutes on day 1. Treatment repeats every 28 days for 4 cycles in the absence of disease progression or unacceptable toxicity. Patients also undergo SBRT on days 36-39 (days 8-11 of cycle 2).
  Interventions: Biological: Anti-CTLA4 Monoclonal Antibody BMS-986218; Radiation: Stereotactic Body Radiation Therapy
- Arm II (BMS-986218, SBRT, nivolumab) (Experimental): Patients receive anti-CTLA4 monoclonal antibody BMS-986218 and SBRT as in Arm 1. Beginning cycle 2, patients also receive nivolumab IV over 30 minutes starting on day 1. Cycles repeat every 28 days for up to 2 years in the absence of disease progression or unacceptable toxicity.
  Interventions: Biological: Anti-CTLA4 Monoclonal Antibody BMS-986218; Biological: Nivolumab; Radiation: Stereotactic Body Radiation Therapy

INTERVENTIONS:
Biological: Anti-CTLA4 Monoclonal Antibody BMS-986218 — Given IV
  Other Names: BMS 986218; BMS-986218; Monoclonal Antibody BMS-986218
Biological: Nivolumab — Given IV
  Other Names: BMS-936558; MDX-1106; NIVO; ONO-4538; Opdivo
  Arms: Arm II (BMS-986218, SBRT, nivolumab)
Radiation: Stereotactic Body Radiation Therapy — Undergo SBRT
  Other Names: SABR; SBRT; Stereotactic Ablative Body Radiation Therapy

SUMMARY:
This phase I/II trial studies the side effects of anti-CTLA4-NF monoclonal antibody (mAb) (BMS986218), nivolumab, and stereotactic body radiation therapy in treating patients with solid malignancies that has spread to other places in the body (metastatic). Immunotherapy with monoclonal antibodies, such as anti-CTLA4-NF mAb (BMS-986218) and nivolumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Stereotactic body radiation therapy uses special equipment to position a patient and deliver radiation to tumors with high precision. This method may kill tumor cells with fewer doses over a shorter period and cause less damage to normal tissue. Giving -CTLA4-NF mAb (BMS986218), nivolumab, and stereotactic body radiation therapy may kill more tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate the safety profile of intravenous anti-CTLA4 monoclonal antibody BMS-986218 (anti-CTLA4-NF mAb [BMS-986218]) alone or with nivolumab administered in combination with stereotactic body radiation therapy (SBRT) targeting 1-4 lesion(s) for patients with metastatic cancers.

SECONDARY OBJECTIVES:

I. To determine antitumor activity of anti-CTLA4-NF mAb (BMS-986218) therapy with SBRT treatment for 1-4 lesions in non-irradiate tumors (abscopal lesions; out of external beam radiation [XRT] field) as defined by Immune-Related Response Criteria (irRC).

II. To determine antitumor activity of anti-CTLA4-NF mAb (BMS-986218) therapy with RadScopal treatment in the low dose treated lesion as defined by irRC.

III. To evaluate treatment efficacy in different SBRT treatment sites (liver versus [vs.] adrenal, lung vs. adrenal).

IV. To evaluate treatment efficacy by comparing anti-CTLA4-NF mAb (BMS-986218) alone with SBRT treatment vs. anti-CTLA4-NF mAb (BMS-986218) in combination with nivolumab and SBRT treatment.

EXPLORATORY OBJECTIVES:

I. To evaluate treatment efficacy by comparing anti-CTLA4-NF mAb (BMS-986218) alone or with SBRT treatment vs. ipilimumab alone or with SBRT treatment (previous trial).

II. To evaluate the associations of tumor-associated and systemic immune biomarkers for therapy with clinical response outcomes and toxicity prediction.

III. To evaluate whether skeletal mass, neutrophil, neutrophil to lymphocyte ratio, and tumor bulk are correlated with clinical outcomes and adverse events.

IV. To evaluate whether tumor kinetics in combination with clinical correlates can help determine treatment response.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I: Patients receive anti-CTLA4 monoclonal antibody BMS-986218 intravenously (IV) over 30 minutes on day 1. Treatment repeats every 28 days for 4 cycles in the absence of disease progression or unacceptable toxicity. Patients also undergo SBRT on days 36-39 (days 8-11 of cycle 2).

ARM II: Patients receive anti-CTLA4 monoclonal antibody BMS-986218 and SBRT as in Arm 1. Beginning cycle 2, patients also receive nivolumab IV over 30 minutes starting on day 1. Cycles repeat every 28 days for up to 2 years in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 30 and 60 days and 6 and 12 months after last cycle of anti-CTLA4 monoclonal antibody BMS-986218.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histological confirmation of solid metastatic cancer with at least one metastatic or primary lesion in the bone, adrenal, liver or lung/chest.
* Patients who have completed prior systemic anti-cancer therapies, an interval of 5 drug half-lives or 4-weeks whichever is shorter, is required, prior to enrollment on study. Note: patients with anaplastic thyroid carcinoma will be waived from this inclusion criteria given the rapid trajectory of their disease. In addition, patients with metastatic castration-resistant prostate cancer (CRPC) will be allowed to continue their maintenance therapy with gonadotropin-releasing hormone (GnRH) analogue agents and supportive bone therapy (e.g., denosumab [XGEVA], zoledronic acid [Zometa]).
* All patients must have at least one metastatic or primary lesion within the bone, lung/chest, liver or adrenal located in an anatomical location amenable to radiation treatment with either 50 Gy in 4 fractions, 60 Gy in 10 fractions, or 30 Gy in 5 fx. Patients may not have more then 80% liver displaced with cancer.
* Repeat radiation in fields previously radiated will be allowed at the discretion of the treating physician
* Age >= 18 years
* Women of childbearing potential (WOCBP) must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of human chorionic gonadotropin) within 24 hours prior to the start of study treatment. Subjects of childbearing potential are those who have not been surgically sterilized or have not been in postmenopausal state. Females in postmenopausal state under the age of 55 years must have a serum follicle stimulating hormone, (FSH) level > 40 mIU/mL to confirm menopause
* Women must not be breastfeeding for the duration of the study and 105 days AFTER completion of study treatment for BMS-986218 monotherapy treatment, 155 days AFTER completion of combination therapy (BMS-986218 + nivolumab) or 5 months AFTER completion of nivolumab maintenance treatment
* WOCBP receiving monotherapy or combination therapy treatment with BMS-986218 must agree to follow instructions for method(s) of contraception or be surgically sterile, or abstain from heterosexual activity for the duration of the study and 105 days AFTER completion of study treatment for BMS-986218 monotherapy treatment, 155 days AFTER completion of combination therapy (BMS-986218 + nivolumab) or 5 months AFTER completion of nivolumab maintenance treatment. WOCBP who are continuously not heterosexually active are exempt from contraceptive requirements, but should still undergo pregnancy testing as described in this section. In the case of male participants, during the course of treatment and 165 days AFTER the end of BMS-986218 monotherapy treatment or 215 days AFTER the end of combination therapy treatment (BMS-986218 + nivolumab) or 7 months AFTER completion of nivolumab maintenance treatment the participant should not father a child (condom use is mandatory, even if vasectomized) or donate sperm. Local laws and regulations may require use of alternative and/or additional contraception methods
* Male participants who are sexually active with WOCBP must agree to follow instructions for methods of contraception during monotherapy treatment with BMS-986218 plus 5 half-lives (75 days) of BMS-986218 plus 90 days for a total of 165 days after the end of BMS-986218 monotherapy treatment or 215 days after the end of combination therapy treatment (BMS-986218 + nivolumab), or 7 months AFTER completion of nivolumab maintenance treatment. In addition, male participants must be willing to refrain from sperm donation during this time
* Investigators shall counsel WOCBP, and male participants who are sexually active with WOCBP, on the importance of pregnancy prevention and the implications of an unexpected pregnancy. Investigators shall advise on the use of highly effective methods of contraception that have a failure rate of < 1% when used consistently and correctly
* Eastern Cooperative Oncology Group (ECOG) performance status 0-1 (Karnofsky > 60%)
* Patients must have normal organ and marrow function as defined below: (use of growth factors or blood transfusion to achieve these requirements is not allowed 2 weeks prior to study enrollment). The blood test for the following analytes will be performed at screening/baseline and at the first day of every BMS-986218 therapy cycle
* Total bilirubin =< 2.0 x upper limit of normal (ULN), except participants with Gilbert's syndrome who must have normal direct bilirubin
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamic pyruvic transaminase [SGPT]) =< 2.5 X institutional upper limit of normal
* Whole blood cell (WBC) >= 2500/uL
* Absolute neutrophil count (ANC) >= 1000/uL
* Platelets >= 75K
* Hemoglobin >= 9 g/dL
* Creatinine =< 1.5 x ULN, or creatinine clearance (CrCl) >= 40 mL/min (measured using the Cockcroft-Gault formula)
* Patients must be willing and able to review, understand, and provide written consent before starting therapy
* Patients with brain metastasis will be included as long as they are free of neurologic symptoms related to metastatic brain lesions and do not require or receive steroid therapy or brain metastasis. We will allow patients with stable brain metastases (no radiographic progression for at least 4 weeks following radiation and/or surgery or 4 weeks of observation), no longer taking steroids for at least 2 weeks prior to first dose of study treatment, and with no new neurological signs and symptoms (clinically and radiographically) for >= 4 weeks to enroll on the protocol
* Patients that have previously progressed on immunotherapy such as ipilimumab, anti-PD-I, anti-PDL-1 or talimogene laherparepvec (T-VEC) will be eligible, but progression on immunotherapy is not required

Exclusion Criteria:

* Patients with active, known, or suspected with autoimmune disorders or those who are at risk for flare of auto-immunity or immune-related diseases
* Participants with well controlled asthma and/or mild allergic rhinitis (seasonal allergies) are eligible
* Participants with the following disease conditions are also eligible:

  * Vitiligo.
  * Type 1 diabetes mellitus.
  * Residual hypothyroidism due to autoimmune condition only requiring hormone replacement.
  * Euthyroid participants with a history of Grave's disease (participants with suspected autoimmune thyroid disorders must be negative for thyroglobulin and thyroid peroxidase antibodies and thyroid stimulating immunoglobulin [Ig] prior to the first dose of study treatment).
  * Psoriasis not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger are permitted to enroll
* Active diverticulitis, intra-abdominal abscess, gastrointestinal (GI) obstruction, abdominal carcinomatosis or other known risk factors for bowel perforation
* Any underlying medical or psychiatric condition, which in the opinion of the Investigator, will make the administration of study drug hazardous or obscure the interpretation of adverse event (AE)s: e.g. a condition associated with frequent diarrhea or chronic skin conditions, recent surgery or colonic biopsy from which the patient has not recovered, or partial endocrine organ deficiencies
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, history of congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Known human immunodeficiency virus (HIV) positive status or with positive test for hepatitis B surface antigen. Patients with hepatitis C antibody (Ab) positive will be considered for enrollment only if quantitative polymerase chain reaction (PCR) is negative
* Any non-oncology vaccine therapy used for prevention of infectious diseases (for up to one month prior to or after any dose of BMS-986218). The use of inactivated seasonal influenza vaccines (e.g., Fluzone), will be permitted on study without restriction
* Concomitant therapy with any of the following: IL-2, interferon or other non-study immunotherapy regimens; cytotoxic chemotherapy; immunosuppressive agents; other investigational therapies; or chronic use of systemic corticosteroids while receiving BMS-986218 (as long as steroid replacement is greater than what is required for physiologic replacement, i.e. in hypothyroidism, adrenal insufficiency)
* History of or current immunodeficiency disease or prior treatment compromising immune function at the discretion of the treating physician
* Prior allogeneic stem cell transplantation or organ allograft
* Patients who were intolerant to previous immuno-oncology (IO) drugs with side effects (grade 4 or greater) that were unable to be resolved with treatment, should be excluded
* Patients that have previously received or progressed on any anti-CTLA4-NF drug
* Absolute lymphocyte count below 0.4 x 10^9/L

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2021-03-29 (Actual); Primary Completion 2027-05-27 (Estimated); Study Completion 2027-05-27 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events | Up to 12 months
  The incidence of clinical and laboratory adverse events will be reported and graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events version 5.0. Adverse events will be reported in frequency tables overall, by intensity, and by relationship. Laboratory values will be reported in shift tables and with summary statistics. Chi-squared or Fisher exact tests will be used to compare safety between two arms. Logistic regression may be used to evaluate the predictive potential of tumor-associated and systemic immune biomarkers for toxicity prediction, and whether skeletal mass, neutrophil, neutrophil to lymphocyte ratio, and tumor bulk are correlated with adverse events.

SECONDARY OUTCOMES:
Tumor response | Up to 12 months
  Will be determined using the Immune Related Response Criteria calculated for each arm with 95% exact confidence intervals. Will evaluate for the % abscopal response, which is defined as the best response rate, summing both complete response (CR) and partial response (PR) patients. This will be a measurement of the non-irradiated lesions. The clinical benefit will be defined as CR+ PR + stable disease (minimum of 6 months from time of enrolment). For patients that have progressive disease at the first treatment study (before re-induction treatment with RadScopal radiation therapy), Immune Related Response Criteria response criteria will be also used to evaluate the responses outside the irradiated tumors. Chi-squared test or Fisher exact test will be used to compare the response rate between two arms and different stereotactic body radiation therapy treatment sites (liver versus [vs.] adrenal, lung vs adrenal).

CONTACTS AND LOCATIONS:
Overall Officials: James Welsh, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

DOCUMENTS (1):
  • Informed Consent Form (2022-05-20): https://cdn.clinicaltrials.gov/large-docs/87/NCT04785287/ICF_000.pdf